CLINICAL TRIAL: NCT00948779
Title: Therapeutic Education About Intake of Oral Solutions of Antibiotics in Children Under 6 Year-old at the Emergency Department in Robert Debré Hospital
Brief Title: Antibiotic Education for Children in an Emergency Care Unit
Acronym: ACHEEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ID RCB 2008-A00892-53
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2012-07

CONDITIONS: Otorhinolaryngologic Diseases; Respiratory Tract Infections; Pyelonephritis; Urinary Tract Infections
Keywords: Patient education; Antibiotic; Child; Respiratory tract infection; Patient satisfaction; Parental knowledge; Adherence
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Respiratory Tract Infections; Pyelonephritis; Urinary Tract Infections; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- antibiotics (Other): antibiotic education for children in an emergency care unit: Patient and family's therapeutic education to improve the use of antibiotics at home.
  Interventions: Other: antibiotic education for children in an emergency care unit
- the antipyretic therapy (Experimental): antibiotic education for children in an emergency care unit: Patient and family's therapeutic education to improve the antipyretic therapy at home.
  Interventions: Other: antibiotic education for children in an emergency care unit

INTERVENTIONS:
Other: antibiotic education for children in an emergency care unit — Educational, Behavioral, and Organizational intervention to improve the use of oral antibiotics in children under 6 years
  Arms: antibiotics
Other: antibiotic education for children in an emergency care unit — Educational, Behavioral and Organizational intervention to improve the antipyretic therapy in children under 6 years.
  Other Names: antibiotic education for children an emergency care unit
  Arms: the antipyretic therapy

SUMMARY:
The purpose of this study is to determine if a patient education in acute condition about the intake of oral solution antibiotic in children under 6 year-old are effective to improve the satisfaction about the therapeutic education, the knowledge about antibiotics among the patients' families and thereby decrease the misuses of antibiotics.

DETAILED DESCRIPTION:
Adherence to antibiotic regimen for common childhood illnesses, such as otitis media and streptococcal pharyngitis, is related to a variety of outcomes such as illness' remission, prevention of recurrent infections, maintaining of cost-effectiveness, and prevention of the growth of antibiotic-resistance. A patient and family 's therapeutic education about the intake of an oral solution of antibiotic should decrease the misuses of antibiotic, improve the family 's knowledge and the satisfaction of the patient and his family. Those factors are related to the understanding and adherence to the antibiotic prescription.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking patients seen at the emergency department and discharged with a diagnosis of bacterial infections (urinary and respiratory tract infections, streptococcal pharyngitis, acute otitis media) requiring 5 to 10 days of an oral solution of antibiotic.
* Under 6 year-old.
* No opposition of the parents to be included in the study.
* Personal health insurance.

Exclusion Criteria:

* Chronic pathology such as: Sickle cell disease, AIDS.
* Parents with insufficient knowledge of French.
* Family not reachable by phone.
* Antibiotic's suspected allergy.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
satisfaction (likert scale) | 15 days

SECONDARY OUTCOMES:
Parent's knowledge | 15 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: François Angoulvant, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Result] Angoulvant F, Rouault A, Prot-Labarthe S, Boizeau P, Skurnik D, Morin L, Mercier JC, Alberti C, Bourdon O. Randomized controlled trial of parent therapeutic education on antibiotics to improve parent satisfaction and attitudes in a pediatric emergency department. PLoS One. 2013 Sep 26;8(9):e75590. doi: 10.1371/journal.pone.0075590. eCollection 2013. PMID 24086581